CLINICAL TRIAL: NCT00675935
Title: Translating Fall Risk Status Into Interventions to Prevent Patient Falls: Falls TIPS (Tailoring Interventions for Patient Safety)
Brief Title: Falls - Tailoring Interventions for Patient Safety
Acronym: Falls TIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Robert Wood Johnson Foundation (Other); Massachusetts General Hospital (Other); North Shore Medical Center (Other)
Responsible Party: Principal Investigator, Patricia C. Dykes, Research Program Director, Center for Patient Safety, Research and Practice, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 62572
Record Dates: First submitted 2008-05-08; First posted 2008-05-12 (Estimated); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Patient Falls
Keywords: Patient falls; fall risk; fall prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): One high-risk medical unit at each hospital will be randomly assigned to receive the fall prevention toolkit
  Interventions: Other: Fall Prevention Tool Kit prototype using a randomized design
- 2 (No Intervention): One high-risk medical unit at each hospital will be randomly assigned to receive usual care as it relates to fall prevention; i.e., receives no intervention.

INTERVENTIONS:
Other: Fall Prevention Tool Kit prototype using a randomized design — Based on the results from Phase 1, Phase 2 and consistent with the literature that suggests that multifaceted, tailored interventions are most effective against inpatient falls, the FPTK prototype will be comprised of two interrelated components 1) The Fall Risk Alert and Communication Plan (translates an individual patient's fall risk assessment into a decision support intervention that communicates fall risk status to team members.) and 2) The Patient Safety Plan of Care PSPOC (translates an individual patient's fall risk assessment into a decision support intervention that creates a tailored evidence-based plan of care). The goal of the FPTK Intervention is to communicate risk status and recommended tailored discipline specific-interventions to prevent falls.
  Other Names: FPTK
  Arms: 1

SUMMARY:
The goal of our project is to prevent patient falls by translating an individual patient's fall risk assessment into a decision support intervention that communicates fall risk status, and creates a tailored evidence-based plan of care that will be accessible to members of the care team to prevent falls.

DETAILED DESCRIPTION:
Patient falls are defined as "patients who experience an unplanned descent to the floor". Patient falls in hospitals are a key safety issue and represent the most frequently reported adverse event in acute care settings. Previous work related to fall risk assessment suggests that a large majority of falls (78%) occur as a result of the presence of physiological risk factors such as confusion, incontinence, poor balance and mobility problems. These falls are considered preventable and as such are classified as iatrogenic.

Phase 1 Specific Aim: To describe the current barriers, facilitators, and methods of fall risk communication in acute care settings (2 academic medical center and 2 community hospital units).

1. What fall risk communication exists within the context of patient care workflow that alerts nurses and other providers (physicians, physical therapists, pharmacists) regarding patients' fall risk status?

   * What should the elements of alerts be at the point of care to support fall risk communication to nurses and other interdisciplinary team members?
   * How should the alert be communicated to professional and paraprofessional providers, patients, and families?
2. What communication of actions to prevent falls exists within the context of patient care workflow that promotes use of a fall prevention plan of care?

   * Based on empirical data to reduce barriers and enhance facilitators, how can information systems be used to create and communicate a tailored evidence-based fall risk patient safety plan of care derived from the nursing fall risk assessment?
   * Based on the C-IC conceptual model, how should the tailored evidence-based fall risk patient safety plan of care be communicated to professional and paraprofessional providers, patients, and families?

Phase 2 Specific Aim: To develop a Fall Prevention Tool Kit (FPTK) prototype that includes 1) The Fall Risk Alert and Communication Plan that translates an individual patient's fall risk assessment into an interdisciplinary fall risk status communication and 2) The Patient Safety Plan of Care (PSPOC), that translates the individual patient's fall risk assessment into a decision support intervention that creates a tailored evidence-based plan of care to be used by professional and paraprofessional providers, patients, and family members across acute care settings.

The FPTK will be developed from fall risk assessment literature, evidence-based fall prevention guidelines and knowledge gained from Phase 1. FPTK components will target common risk communication/fall intervention requirements identified in Phase 1 across the four hospitals to facilitate testing the prototype in Phase 3 and to improve generalizability of our findings.

Phase 3 Specific Aim: To evaluate the effectiveness of the FPTK prototype on reducing patient falls.

1. Is the FPTK used to communicate fall risk status and facilitate adherence with the tailored patient safety plan of care recommendations?
2. Is there a relationship between use of the FPTK and the incidence of falls (primary outcome measure) and fall-related injury (secondary outcome measure)?
3. Is there a difference in the frequency with which tailored fall prevention interventions are documented when professional and paraprofessional providers, patients and family members have access to the FPTK when compared to usual care?

Phase 4 Specific Aim: To evaluate satisfaction with the FPTK prototype and to generate recommendations for improvement.

1. Are the interdisciplinary team members, paraprofessionals, patients and family members satisfied with the FPTK?
2. What components are most useful and what recommendations can be made to improve the perceived usefulness and ease of use of the FPTK? If the FPTK works, then one will see that: 1) the tool kit is used and those helpful and useful components will be identified, 2) those who use the tool kit are satisfied with its use, 3) there is a decrease in the incidence of falls and falls with injury.

ELIGIBILITY:
Inclusion Criteria:

* 2 units per hospital for participation. One unit will be randomized to receive the intervention; the other will serve as a control. Inclusion Criteria: Non-specialty (medical) units and units with similar types of patients and fall rates (fall rates higher than hospital mean).
* Identify focus group/interview participants. Interdisciplinary staff members. Selection criteria: nurses, nursing assistants and other providers (12 total more heavily weighted w/nursing staff) to participate in the study focus groups.
* Patients who have fallen (4 patients at each hospital) for participation in phone interview.
* Patients for analysis must be adults admitted to intervention units.

Exclusion Criteria:

* Anyone who does not meet criteria above.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10264 (Actual)
Dates: Start 2007-09; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The outcome measure will be rate of patients falls per 1000 patient days | 1/2009-6/2009
  Specific Aim: To evaluate the effectiveness of the FPTK prototype on reducing patient falls.
  1. Is the FPTK used to communicate fall risk status and facilitate adherence with the tailored patient safety plan of care recommendations?
  2. Is there a relationship between use of the FPTK and the incidence of falls (primary outcome measure)?

SECONDARY OUTCOMES:
Falls with injury as a secondary outcome measure. | 1/2009-6/2009
  Is there a relationship between use of the FPTK and the incidence of Fall-related injury (secondary outcome measure)
To evaluate the effectiveness of the FPTK prototype on documentation of planned and completed tailored interventions | 1/2009-6/2009
  Is there a difference in the frequency with which tailored fall prevention interventions are documented when professional and paraprofessional providers, patients and family members have access to the FPTK when compared to usual care?

CONTACTS AND LOCATIONS:
Overall Officials: Lana Tsurikova, MSc, MA, Study Director — Partners Healthcare Sys; Patricia C. Dykes, RN, DNSc, Principal Investigator — Partners Healthcare Sys
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

REFERENCES:
- [Derived] Dykes PC, Carroll DL, Hurley A, Lipsitz S, Benoit A, Chang F, Meltzer S, Tsurikova R, Zuyov L, Middleton B. Fall prevention in acute care hospitals: a randomized trial. JAMA. 2010 Nov 3;304(17):1912-8. doi: 10.1001/jama.2010.1567. PMID 21045097